CLINICAL TRIAL: NCT02228330
Title: Prospective Clinical Trial - Obturator Reflex Predictors and Blockage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0063-14-RMC
Record Dates: First submitted 2014-08-04; First posted 2014-08-29 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Malignant Neoplasm of Urinary Bladder
Keywords: Transurethral resection of bladder tumors; Obturator nerve reflex; Obturator nerve block
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- uni-lateral obturator nerve block (Experimental): Patients scheduled for TUR for bladder tumor Intervention: uni-lateral obturator nerve block.
  non-blocked obtorator side of each patient will be used as control
  Interventions: Procedure: obturator nerve block

INTERVENTIONS:
Procedure: obturator nerve block — a uni-lateral obturator nerve block will be performed under ultrasound guidance- using 2% lidocaine for obtaining a short term block.

SUMMARY:
The aim of this study is to estimate the incidence rate of obturator nerve reflex and leg jerking during Transurethral Resections of Bladder Tumors (TURBTs), evaluate the efficacy of obturator nerve block in the prevention of inadvertent muscle spasm, and to identify predictors for both the jerking reflex and successful nerve block.

DETAILED DESCRIPTION:
Study design: A single center single arm prospective study aiming to estimate the incidence rate of obturator nerve reflex and leg jerking during TURBTs, evaluate the efficacy of obturator nerve block (ONB) in the prevention of inadvertent muscle spasm, and identify predictors for both the jerking reflex and successful nerve block.

Study population: patients who are scheduled for TUR for bladder tumor, as standard care, who are willing and able to participate in the study

Intervention: a uni-lateral ONB (using Lidocaine 2%)

Study outline: Once in the operating room patients will be monitored by continuous electrocardiography, non-invasive arterial blood pressure measurement, and pulse oximetry in the usual manner. They will then undergo general or spinal anesthesia according to their preference and at the discretion of the treating anesthesiologist, without the use of muscle relaxants. As part of the study, a uni-lateral ONB will be performed under ultrasound guidance- using 2% lidocaine for obtaining a short term block, for the duration of the procedure itself. The non-blocked nerve will be used as control. The surgeon will be blinded as to the side in which the ONB has been performed. A catheter will be used to fill the bladder with saline to its full capacity. The inner wall of the bladder will then be stimulated to test for an obturator nerve reflex and leg jerking. Stimulation will be done using a trans-resectoscope and a single-twitch electrical current generated by a neuromuscular monitoring device, as previously described by Mihara et al. Four different bladder volumes will be tested. For each bladder volume, a reflex response on both sides will be documented and graded. The investigators will then proceed with a TUR in the usual manner.

Primary endpoints: frequency of obturator jerk reflex and efficacy of obturator nerve block

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, older than 18 yo, scheduled for TUR for bladder tumor.
* The subject is willing and able to read, understand and sign the study specific informed consent form.

Exclusion Criteria:

* Patients with known coagulopathy, including patients receiving antithrombotic or thrombolytic therapy not in compliance with standard precautions.
* Patients with a known allergy to anesthetics.
* Patients who underwent partial cystectomy.
* Patients with tumors involving bladder diverticula.
* Patients with pre-existing obturator nerve injury or pre-existing neurologic deficits.
* Patients with neuromuscular disease.
* Patients with local infection above planned ONB site.
* Patients in whom the use of muscle relaxants is deemed necessary by the anesthesiologist.
* Patients with inguinal lymphadenopathy.
* Patients unable to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
efficacy of obturator nerve block in preventing inadvertent obturator jerk | intraoperative
  percentage of subjects for which the obtorator nerve block prevnted inadvertent obturator jerk

SECONDARY OUTCOMES:
incidence rate of obturator nerve jerk reflex | end of study (one year)
  frequency of obturator nerve jerk reflex

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD, PhD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided